CLINICAL TRIAL: NCT03221712
Title: The Registry Study to Compare the Cardiopulmonary Exercise Test Parameters Before and After Cardiac Rehabilitation in Patients With Chronic Total Occlusion of the Coronary Arteries
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV retrospective
Record Dates: First submitted 2017-07-16; First posted 2017-07-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Coronary Artery Disease; Total Occlusion of Coronary Artery
Keywords: cardiopulmonary exercise test; chronic total occlusion; cardiac rehabilitation
MeSH Terms: conditions — Coronary Artery Disease | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: cardiac rehabilitation — cardiac rehabilitation in patients with chronic total occlusion of the coronary arteries.

SUMMARY:
The aim of this study is to find strategy for treatment through comparing the cardiopulmonary exercise test parameters before and after cardiac rehabilitation in patients with chronic total occlusion of the coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and more
* Chronic total occlusion of coronary artery disease
* Cardiac rehabilitation

Exclusion Criteria:

* Not applicable

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac rehabilitation in patients with chronic total occlusion of the coronary arteries.
Sampling Method: Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Death | 5 year
Myocardial infarction | 5 year
Repeat revascularization | 5 year

SECONDARY OUTCOMES:
Maximum rate of oxygen consumption | 5 year
  maximum rate of oxygen consumption as measured during incremental exercise, most typically on a motorized treadmill.
Respiratory exchange ratio | 5 year
Maximal heart rate | 5 year
Physical activity_METs | 5 year
  Physical activity is measured in metabolic equivalents (METs), which are multiples of the resting rate of O2 consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided